CLINICAL TRIAL: NCT01455402
Title: An Observational Study to Assess Respiratory Syncytial Virus (RSV)-Associated Illness in Adults With Chronic Obstructive Pulmonary Disease (COPD) and/or Congestive Heart Failure (CHF)
Brief Title: An Observational Study to Assess RSV-associated Illness in Adults With COPD and/or CHF
Acronym: CD-1089
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-ID-MEDI-557-1089; D3150L00001 (Other: AstraZeneca AB)
Record Dates: First submitted 2011-10-12; First posted 2011-10-20 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Syncytial Virus, Chronic Obstructive Pulmonary Disease, Congestive Heart Failure
Keywords: Respiratory Syncytial Virus, Chronic Obstructive Pulmonary Disease, Congestive Heart Failure, Observational
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, whole blood, plasma, nasal swab, sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this observational study is to determine the incidence of medically attended (inpatient or outpatient) acute respiratory illnesses or events leading to worsening cardiorespiratory status (ie, acute exacerbations of chronic obstructive pulmonary disease [AECOPD] or worsening CHF) associated with RSV infections in high-risk adults (ie, those with severe COPD and/or advanced CHF) across multiple consecutive RSV seasons.

DETAILED DESCRIPTION:
It is expected that this observational study will provide further understanding of the clinical impact and true incidence rates of RSV-associated hospitalizations and medically attended acute respiratory illnesses or events leading to worsening cardiorespiratory status in adults with COPD and/or CHF who are at increased risk for serious sequelae associated with RSV infections. As part of the evaluation, this study will collect symptom and physiologic data, and blood, nasal swab, and sputum in order to investigate the relationship of RSV infections with clinical endpoints.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 50 years or greater
* Hospitalization due to worsening COPD and/or CHF
* Severe COPD subjects (Global Initiative for Obstructive Lung Disease Stage III/IV); FEV1 <50%
* Chronic CHF subjects (New York Heart Association Class III/IV or American College of Cardiology-American Heart Association Stage C/D); Ejection fraction < 40%
* Expects to have direct contact with children at least once a month

Key Exclusion Criteria:

- Participation in another clinical study involving the use of investigational product

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults with severe COPD and/or CHF who expect to have contact with children. Potential subjects will be identified through the medical record and extended invitations to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incidence rate of inpatient RSV-associated acute respiratory illness or events leading to worsening cardiorespiratory status | Average of 2 years

SECONDARY OUTCOMES:
All-cause inpatient acute respiratory illnesses or events leading to worsening cardiorespiratory status | Average of 2 years
Mortality through all RSV seasons of follow up for RSV-associated deaths and all-cause deaths | Average of 2 years
Healthcare utilization for RSV-associated and all-cause medically attended acute respiratory illnesses or events leading to worsening cardiorespiratory status | Average of 2 years
Incidence of RSV-associated secondary bacterial pneumonia events | Average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pam Griffin, MD, Study Director — MedImmune LLC
Locations (54):
- United States (21):
  - Research Site, Birmingham, Alabama
  - Research Site, Fort Smith, Arkansas
  - Research Site, Denver, Colorado
  - Research Site, Bay Pines, Florida
  - Research Site, Miami, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Council Bluffs, Iowa
  - Research Site, Minneapolis, Minnesota
  - Research Site, Reno, Nevada
  - Research Site, Buffalo, New York
  - Research Site, Mineola, New York
  - Research Site, Rochester, New York
  - Research Site, Chardon, Ohio
  - Research Site, Beaver, Pennsylvania
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Marshfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Bulgaria (3):
  - Research Site, Pleven, Pleven
  - Research Site, Razgrad, Razgrad
  - Research Site, Sofia, Sofia
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint Romuald, Quebec
- Czechia (5):
  - Research Site, Jindrichuv Hradec III
  - Research Site, Kyjov
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Rokycany
- France (3):
  - Research Site, Lyon, France
  - Research Site, Toulouse, France
  - Research Site, Nantes
- Germany (3):
  - Research Site, Berlin
  - Research Site, Leipzig
  - Research Site, Mannheim
- Italy (5):
  - Research Site, Ferrara, FE
  - Research Site, Florence, FI
  - Research Site, Genova, GE
  - Research Site, Pisa, PI
  - Research Site, Parma, PR
- Russia (2):
  - Research Site, Moscow
  - Research Site, Novosibirsk
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Uppsala